CLINICAL TRIAL: NCT05998915
Title: A Multi-center Study on Human Microecology Assisted Diagnosis of Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CALM2102
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-03

CONDITIONS: Human Microecology；Colorectal Disease；Auxiliary Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Colorectal Cancer(CRC): People who is diagnosed with CRC by colonoscopy and pathological biopsy
  Interventions: Other: observe only
- Inflammatory Bowel Disease: People who is diagnosed with IBD by colonoscopy and pathological biopsy
  Interventions: Other: observe only
- Colorectal adenoma(CRA)/adenomatous polyposis: People who is diagnosed with CRA by colonoscopy and pathological biopsy
  Interventions: Other: observe only
- Non-adenomatous polyps: People who is diagnosed with non-adenomatous polyps by colonoscopy and pathological biopsy
  Interventions: Other: observe only
- Irritable bowel syndrome: People who is diagnosed with IBS by colonoscopy and pathological biopsy
  Interventions: Other: observe only
- normal: People who has no obvious abnormality in the whole colon
  Interventions: Other: observe only

INTERVENTIONS:
Other: observe only — observe only

SUMMARY:
As for this research，we want to find whether the intestinal microecology (flora, peptidoglycan fragments) have certain distribution characteristics in colorectal diseases; whether it can predict the development of disease/as a prognostic indicator.

DETAILED DESCRIPTION:
We even want to find whether it can predict the development of disease/as a prognostic indicator.

ELIGIBILITY:
Inclusion Criteria:

* people who is going to get the colonoscopy examination

Exclusion Criteria:

* people who was diagnosed as one cancer，expect for CRC; who has had the antibiotics or the medicine that treats for colorectal disease, except for medical probiotics, in one month; who has had the laxative and the colonscopy in one week; who had a operation in three month.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 2500
Sampling Method: Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
collect specimen before colonscope | Baseline (before colonscope)
  collect fecal，saliva，urine，blood to assess the level of the activation of NOD2，cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China